CLINICAL TRIAL: NCT06888037
Title: A Prospective, Multicenter Clinical Study of Fruquintinib Combined With PD-1 Monoclonal Antibody as First-line Maintenance Therapy in Patients With HER-2-negative Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Fruquintinib Combined With PD-1 Inhibitor as First-line Maintenance Therapy for Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-G114
Record Dates: First submitted 2025-03-12; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Gastric Adenocarcinoma; GEJ Adenocarcinoma; First-line Therapy; Maintenance Therapy; Fruquintinib; PD-1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: fruquintinib＋PD-1 (maintenance treatment) (Experimental)
  Interventions: Drug: Initial treatment: PD-1+ Oxaliplatin-based chemotherapy (CAPOX/SOX/FOLFOX）; Drug: Maintenance treatment (after 3 months): fruquintinib+PD-1

INTERVENTIONS:
Drug: Initial treatment: PD-1+ Oxaliplatin-based chemotherapy (CAPOX/SOX/FOLFOX） — CAPOX/SOX (each cycle is 21 days): Oxaliplatin 130mg/m2, ivgtt, D1; Capecitabine 1000 mg/m2, po, bid, D1-14 or S-1: 40-60mg according to BSA, bid, D1-14.
  FOLFOX (each cycle is 14 days): Oxaliplatin 85mg/m2, ivgtt, D1, Q2W; 5-Fluorouracil: 400mg/m2, D1, followed by 2400 mg/m2 as a continuous IV infusion over 46 hours; Leucovorin: 400mg/m2, iv, D1.
  PD-1 monoclonal antibody:
  Nivolumab 360mg/3 weeks or 240mg /2 weeks, iv, D1; If weight ≥60 kg, Sintilimab 200mg/3 weeks; if weight < 60 kg, Sintilimab 3mg/kg/3 weeks, iv, D1; Tislelizumab 200mg/3 weeks, iv, D1; Pembrolizumab 200mg/3 weeks, iv, D1;
Drug: Maintenance treatment (after 3 months): fruquintinib+PD-1 — After 3 months (12 weeks) of initial treatment with oxaliplatin-based chemotherapy combined with PD-1 monoclonal antibody, those with complete response (CR), partial response (PR) or stable disease (SD) assessed by imaging evaluation continued to receive maintenance treatment with furoquininib and PD-1 monoclonal antibody.
  Fruquintinib 3 mg/d, qd po, D1-21, Q4W; PD-1 monoclonal antibody is repeated as initial treatment until the disease progresses or unacceptable toxicity.

SUMMARY:
This study was designed to explore the efficacy and safety of fruquintinib combined with PD-1 inhibitors as first-line maintenance therapy for advanced HER-2 Negative Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed the informed consent and had good compliance;
* Age ≥18 years, Eastern Cooperative Oncology Group (ECOG) score 0-1, and expected survival time ≥12 months;
* Histologically or cytologically unresectable, locally advanced, recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma;
* He had not received previous systemic chemotherapy for unresectable, locally advanced, recurrent, or metastatic gastric or gastroesophageal junction adenocarcinoma;
* Patients with disease progression/relapse occurring more than 6 months after completion of neoadjuvant/adjuvant therapy;
* At least one measurable lesion according to RECIST version 1.1;
* Tumor tissue/serum samples were tested as microsatellite stable (MSS) or mismatch repair intact (pMMR), HER2 negative;
* Adequate organ functions:

Absolute neutrophil count ≥1.5×109/L; Platelet ≥100×109/L; Hemoglobin ≥90g/L; WBC≥3×109/L Total bilirubin ≤ 1.5XULN; ALT and AST ≤2.5XULN (If liver metastasis, AST and ALT≤5 XULN)； Serum creatinine (Cr) ≤1.5XULN or serum creatinine clearance ≥50 ml/min； Urinary protein ≤2+, or 24-hour urinary protein volume ≤2000mg; Prothrombin time (PT) and partially activated prothrombin time (APTT) ≤1.5×ULN;

• Female or male patients of reproductive age must use effective contraception throughout and for 6 months after treatment.

Exclusion Criteria:

* Participated in other drug clinical trials within 4 weeks before enrollment;
* Have had other malignancies within the past 5 years, except cured basal cell carcinoma of the skin, papillary carcinoma of the thyroid, superficial bladder, carcinoma in situ of the breast, and carcinoma in situ of the cervix ;
* History of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥ grade 2 (NCI-CTCAE 5.0), heart failure ≥ grade 2 New York Heart Association (NYHA), transmural myocardial infarction, unstable angina, poorly controlled arrhythmia, etc.
* Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) and type 2 diabetes uncontrolled by antidiabetic treatment (fasting blood glucose ≥8.9mmol/L);
* Active autoimmune and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease, and Hashimoto's thyroiditis;
* Type 1 diabetes mellitus, hypothyroidism that can be controlled only with replacement therapy, and skin diseases (e.g., vitiligo, psoriasis) that do not require systemic treatment could be included;
* Central nervous system (CNS) metastases that are not adequately treated, or the presence of uncontrolled or symptomatic active CNS metastases; Patients with adequately treated CNS metastases and neurologic symptoms that had returned to baseline at least 4 weeks before enrollment (with the exception of residual signs or symptoms related to CNS therapy) were eligible for enrollment; In addition, participants had to discontinue corticosteroids or to be taking a stable or tapering dose of prednisone (or equivalent doses of other corticosteroids) of 10 mg or less per day at least 4 weeks before enrollment;
* The patients had pleural effusion and ascites that could not be controlled by puncture drainage and other treatments within 14 days before enrollment. Moderate or greater pericardial effusion with clinical symptoms;
* A live or attenuated live vaccine was administered within 30 days before enrollment;
* Major surgery had been performed within 28 days before enrollment or minor nonstudy-related surgery had been performed within 7 days before enrollment (with the exception of tumor biopsy and venous-access port placement);
* Patients with clinically significant bleeding symptoms or definite bleeding tendency within 3 months before enrollment; Patients with gastrointestinal perforation and/or gastrointestinal fistula within 6 months before enrollment (except those whose symptoms disappeared after gastric cancer resection for bleeding/perforation of gastric cancer);
* Arterial/venous thrombotic events, such as cerebrovascular accident (including transient ischemic attack, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months beforeenrollment;
* Major vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral thrombosis) within 6 months before enrollment;
* Severe, unhealed or open wounds and active ulcers or untreated fractures;
* Had a history of immediate anaphylaxis;
* The presence of clinically significant pulmonary fibrosis or interstitial pneumonia as judged by the investigator; Had active lung infection prior to injection and required anti-infective therapy;
* Active infections included tuberculosis (medical history, investigator's judgment, radiological examination, and local laboratory testing), hepatitis B (hepatitis B surface antigen positive and HBV DNA above the upper limit of the study center's normal range), hepatitis C (HCV antibody positive and HVC RNA positive), HIV (HIV antibody positive), syphilis, etc;
* Had active gastrointestinal bleeding or hemoptysis;
* A history of alcohol or psychotropic substance abuse with no withdrawal or a history of mental disorder;
* Known allergy to the study drug or any of its excipients; Or severe allergic reactions to other monoclonal antibodies;
* Systemic antibiotic use for ≥ 7 days within 4 weeks before enrollment or unexplained fever >38.5°C during screening or before the first dose (fever due to a neoplastic cause, as judged by the investigator, was eligible);
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Unable to take oral medication;
* The presence of other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the results of the study, and patients who were deemed by the investigators to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year progression-free survival rate | Up to 1 year
  The proportion of patients who remain alive and free from disease progression for at least 12 months after initiating treatment.

SECONDARY OUTCOMES:
One-year overall survival rate | Up to 1 year
  The proportion of patients who remain alive for at least 12 months after initiating treatment.
Two-year overall survival rate: | Up to 2 years
  The proportion of patients who remain alive for at least 24 months after initiating treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided